CLINICAL TRIAL: NCT06099418
Title: A Two-Arm Randomized, Double-Blind, Placebo-Controlled Phase 2 Selection Trial to Evaluate the Efficacy and Safety of VB10.16 Alone or in Combination With Atezolizumab in Patients With HPV16-Positive, PD-L1-positive, Recurrent or Metastatic Cervical Cancer Who Are Refractory to Pembrolizumab With Chemotherapy With/Without Bevacizumab.
Brief Title: Efficacy and Safety of VB10.16 Alone or in Combination With Atezolizumab in Patients With Advanced Cervical Cancer.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial VB-C-04 was stopped due to company strategic reasons and recent changes in standard of care in the recurrent and metastatic cervical cancer setting.
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Roche Pharma AG (Industry); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB-C-04; GOG-3091 (Other: GOG Foundation)
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: HPV-Related Cervical Carcinoma; HPV-Related Malignancy; Cervical Cancer
Keywords: Recurrent; metastatic; HPV16-positive; PD-L1 positive
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence; Neoplasm Metastasis | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: A modified randomized phase 2 selection ('pick-the-winner') design with a margin of practical equivalence will be implemented to monitor efficacy of the two individual arms, and to decide which of the two arms that may be continued further based on the primary endpoint of confirmed ORR.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VB10.16 + placebo (Experimental): 9 mg VB10.16 via i.m. needle free injections in the deltoid muscles and quadricep or gluteus muscle.
  Placebo will be given via IV infusions.
  Interventions: Biological: VB10.16; Drug: Placebo
- VB10.16 + atezolizumab (Experimental): 9 mg VB10.16 via i.m. needle free injections in the deltoid muscles and quadricep or gluteus muscle.
  Atezolizumab will be given via IV infusions.
  Interventions: Biological: VB10.16; Drug: Atezolizumab Injection [Tecentriq]

INTERVENTIONS:
Biological: VB10.16 — Intramuscular (i.m.) administrations of VB10.16 every 3 weeks (Q3W) during a 12-week induction period, followed by a maintenance period with administrations every 6 weeks (Q6W) from Week 13 until Week 49.
  A total of up to 11 i.m. administrations will be given. VB10.16 will be administered via Pharma Jet® Stratis 0.5 mL needle free injection system.
Drug: Atezolizumab Injection [Tecentriq] — Intravenous (IV) infusions of atezolizumab (saline solution) every 3 weeks.
  Arms: VB10.16 + atezolizumab
Drug: Placebo — Intravenous (IV) infusions of placebo (saline solution) every 3 weeks.
  Arms: VB10.16 + placebo

SUMMARY:
This is a multi-center study in patients with recurrent or metastatic HPV16-positive, PD-L1 positive cervical cancer who has progressed during or after treatment with the first-line standard of care (pembrolizumab with chemotherapy with/without bevacizumab).

The trial is designed to investigate VB10.16 alone or in combination with the immune checkpoint inhibitor, atezolizumab.

The trial consist of 2 parts: the first part which investigates VB10.16 + placebo versus VB10.16 + atezolizumab. Approximately 30 patients will be included in each group. The goal of this part is to evaluate which of the two treatments is the best.

The second part of the study will select the best treatment from part 1 and investigate the safety and efficacy of additional 70 patients.

DETAILED DESCRIPTION:
This is a two-arm randomized, double-blind, placebo-controlled phase 2 selection trial to evaluate the efficacy and safety of VB10.16 alone or in combination with atezolizumab in patients with HPV16-positive, PD-L1-positive, recurrent or metastatic cervical cancer who are refractory to pembrolizumab with chemotherapy with/without bevacizumab. A selection design with a margin of practical equivalence will be implemented to monitor efficacy of the two experimental arms (VB10.16 + atezolizumab vs. VB10.16 + placebo).

The trial consist of 2 parts: the first part which investigates VB10.16 + placebo versus VB10.16 + atezolizumab. Approximately 30 patients will be included in each group. The goal of this part is to evaluate which of the two treatments is the superior.

The second part of the study will select the superior treatment from part 1 and investigate the safety and efficacy of additional 70 patients.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years at ICF signature date.
2. Persistent recurrent or metastatic (R/M) (stage IVB) PD-L1 positive cervical cancer with squamous cell, adenocarcinoma or adenosquamous histology with confirmed disease progression during or after treatment with 1st line systemic standard of care pembrolizumab + platinum-containing chemotherapy +/- bevacizumab

   1. Participants should have received at least 4 cycles of pembrolizumab.
   2. Planned treatment start should be within 12 weeks of documented radiographic disease progression.
   3. Participants should have received no more than 1 prior systemic anti-cancer treatment regimen for recurrent/metastatic cervical cancer (pembrolizumab + chemotherapy +/- bevacizumab).
3. PD-L1-positive tumor confirmed by Ventana SP263 clone (the Food and Drug Administration approved companion diagnostic test for atezolizumab in other indications), with tumor area positivity ≥5% in designated central laboratory
4. HPV16-positive tumor confirmed by nucleic acid amplification test in designated central laboratory
5. At least 1 measurable lesion per RECIST v1.1 as assessed by Blinded Independent Central Review.

   Overall function and organ function:
6. ECOG performance status (PS) ≤1
7. Gustave Roussy Immune (GRIm) score ≤1

Key Exclusion Criteria:

Disease specific:

1. Has disease that is suitable for local therapy with curative intent.
2. Rapidly progressing disease (e.g., tumor bleeding, uncontrolled tumor pain) in the opinion of the investigator.
3. Neuroendocrine carcinoma of the cervix.

   Prior, concurrent or future interventions:
4. Radiotherapy (or other non-systemic therapy) ≤14 days prior to VB10.16 treatment start, or the patient has not fully recovered (i.e., Grade ≤1 at baseline) from AEs due to a previously administered treatment.
5. Has received prior surgery or prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment.
6. Prior solid organ or tissue transplantation (except corneal transplant).
7. Prior autologous or allogeneic hematopoietic stem cell transplantation.
8. Prior chimeric antigen receptor T-cell (CAR-T) therapy.
9. Prior therapy with a monoclonal antibody, bispecific antibody, or antibody fragment (or other molecule with similar mechanism of action) that engages with stimulatory or co-inhibitory molecules on T cells (e.g., CD3, CTLA-4, PD-1, 4-1BB/CD137), except pembrolizumab in the metastatic setting.
10. Prior therapy with CPI in the locally advanced setting.
11. Prior administration with tisotumab vedotin.
12. Administration of a live (attenuated replicating organism) or non-live (pathogen component or killed whole organism) vaccine, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine within 30 days prior to VB10.16 treatment start.
13. Prior administration with a therapeutic HPV16 vaccine.
14. Prior severe hypersensitivity (≥ grade 3) to atezolizumab and/or any of its excipients.
15. Prior persistent toxicities (≥ grade 3) related to pembrolizumab administration.
16. Participants receiving systemic immunosuppression with immunosuppressive agents such as cyclosporine, azathioprine, methotrexate, or tumor necrosis factor alpha blockers for any concurrent condition.
17. Chronic administration of systemic corticosteroids: prednisone >10 mg daily (or dose equivalent) or an average cumulative dose of >140 mg prednisone (or dose equivalent) within the last 14 consecutive days prior to VB10.16 treatment start.
18. Any planned major surgery.

    Prior or concurrent morbidity:

    Malignancy:
19. Past or current malignancy other than inclusion diagnosis, except for:

    1. Noninvasive basal cell or squamous cell skin carcinoma.
    2. Noninvasive, superficial bladder cancer.
    3. Ductal carcinoma in situ.
    4. Any curable cancer with a complete response of >2 years' duration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 1 year
  Objective Response Rate (ORR), defined as the proportion of patients who have either confirmed CR or confirmed PR as best overall response per RECIST 1.1 as assessed by blinded independent central review (BICR).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 year
  Objective Response Rate (ORR), defined as the proportion of patients who have either confirmed CR or confirmed PR as best overall response per RECIST 1.1 as assessed by the investigator.
Duration of Response (DOR) | Up to approximately 2 years
  Duration of response (DOR) based upon RECIST v1.1 assessed by BICR. DOR is defined as time from the date of first documented response of confirmed CR or PR to the date of the first documented progression or death due to any cause, whichever occur first.
Duration of Response (DOR) | Up to approximately 2 years
  Duration of response (DOR) based upon RECIST v1.1 assessed by the investigator. DOR is defined as time from the date of first documented response of confirmed CR or PR to the date of the first documented progression or death due to any cause, whichever occur first.
Time to Response (TTR) | Up to approximately 2 years
  Time to response (TTR) based upon RECIST v1.1 assessed by BICR. TTR is defined as the time from VB10.16 treatment start date to the date of first documented response of either confirmed CR or confirmed PR.
Disease Control Rate (DCR) | Up to approximately 2 years
  Disease Control Rate (DCR) based upon RECIST v1.1 assessed by BICR. DCR is defined as the proportion of patients who have either confirmed CR, confirmed PR, or SD as best overall response.
Duration of Disease Control (DODC) | Up to approximately 2 years
  Duration of disease control (DODC) based upon RECIST v1.1 assessed by BICR. DODC is defined as time from the date of first documented response of confirmed CR, confirmed PR or SD to the date of the first documented progression or death due to any cause.
Progression Free Survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) as assessed by BICR. PFS is defined as the time from the VB10.16 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Progression Free Survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) as assessed by the investigator. PFS is defined as the time from the VB10.16 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 2 years
  Overall survival (OS), defined as the time from VB10.16 treatment start date to the date of death from any cause.
Minimal Response | Up to approximately 2 years
  Proportion of participants with tumor shrinkage ≥10.0% to <30% assessed by BICR.
Proportion of participants who are Progression-free | 26 weeks
  Proportion of participants who are progression-free and alive based upon RECIST v1.1 assessed by BICR.
Proportion of participants who are Progression-free | 52 weeks
  Proportion of participants who are progression-free and alive based upon RECIST v1.1 assessed by BICR.
Proportion of participants who are Progression-free | 104 weeks
  Proportion of participants who are progression-free and alive based upon RECIST v1.1 assessed by BICR.
Proportion of participants who are alive. | 26 weeks
  Proportion of participants who are alive.
Proportion of participants who are alive. | 52 weeks
  Proportion of participants who are alive.
Proportion of participants who are alive. | 104 weeks
  Proportion of participants who are alive.
Molecular Response | Up to week 52
  Proportion of participants with molecular response defined as ≥30% decrease from baseline in HPV16 ctDNA.
Molecular Response | Up to week 52
  Proportion of participants with molecular response defined as ≥50% decrease from baseline in HPV16 ctDNA.
Proportion of participants with treatment emergent adverse events | Up to week 104
  Proportion of participants with treatment-emergent adverse events (TEAEs) by severity grade.
Proportion of participants with treatment-emergent serious adverse events | Up to week 104
  Proportion of participants with treatment-emergent serious adverse events
Proportion of participants with drug related toxicity | Up to week 104
  Proportion of participants with drug-related toxicity of CTCAE grade ≥3
Proportion of participants with discontinuation | Up to week 104
  Proportion of participants discontinuing treatment due to an adverse reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Salani, MD MBA, Principal Investigator — UCLA Division of Gynecologic Oncology

IPD SHARING:
Plan to Share IPD: No